CLINICAL TRIAL: NCT05617846
Title: Efficacy and Safety of Antiosteoporosis Therapy in Patients After Bone Tumor Resection: a Multicenter, Real-world Prospective Cohort Observational Study
Brief Title: Application of Antiosteoporosis Therapy in Osteolysis
Status: Not yet recruiting | Type: Observational
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Wang Jiaqiang, associate chief physician, Henan Cancer Hospital
Other Study IDs: ZZUSC-19
Record Dates: First submitted 2022-10-31; First posted 2022-11-16 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2023-08

CONDITIONS: Limb; Fusion; Complication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention group: Patients who received antiosteoporosis therapy after bone tumor resection
  Interventions: Other: Anti-osteoporosis therapy
- Control group: Patients who underwent bone tumor resection without antiosteoporosis therapy

INTERVENTIONS:
Other: Anti-osteoporosis therapy — Bone healing, limb function, and complications of postoperative osteolysis in patients with bone tumors of the extremities treated with anti-osteoporosis therapy.
  Groups: Intervention group

SUMMARY:
To report the postoperative complications and limb function of patients with osteolysis after surgery for bone tumors of the extremities who received anti-osteoporosis therapy in Henan Cancer Hospital in the next 10 years.

DETAILED DESCRIPTION:
A total of 100 patients with osteolysis after surgery for bone tumors of the four extremities who received anti-osteoporosis treatment in Henan Cancer Hospital in the next 10 years were reported. The basic information, treatment methods, postoperative complications and limb function of these patients were collected.

ELIGIBILITY:
Inclusion Criteria:

1. No age restriction, male or female.
2. A subtype of bone tumor (including benign, malignant, and metastatic cancer) was confirmed in the pathology department of the research institution.
3. Received excision of bone tumor in research institution.

Exclusion Criteria:

Not applicable.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving antiosteoporosis therapy for osteolysis after surgery for bone tumors in the extremities
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-28 (Estimated); Primary Completion 2032-11-30 (Estimated); Study Completion 2032-11-30 (Estimated)

PRIMARY OUTCOMES:
Complications | Collected from the beginning of treatment to 24 months after treatment.
  The incidence of complications after anti-osteoporosis treatment was collected and the severity of complications was evaluated according to CTCAE5.0.
Limb function | Collected from the beginning of treatment to 24 months after treatment.
  Limb function was assessed using the Musculoskeletal Oncology Society (MSTS) scoring scale for seven items, namely movement, pain, stability, deformity, strength, functional activity, and emotional receptiveness. The highest possible score is 35, with 5 points allocated to each project.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Bone and Soft Tissue ,Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No